CLINICAL TRIAL: NCT04763564
Title: Efficacy of Liraglutide Therapy in Patients With an Ileal -Pouch Anal Anastomosis (IPAA) and Chronic High Bowel Frequency
Brief Title: Efficacy of Liraglutide Therapy in Patients With IPAA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to an interruption in drug supply, the study was terminated
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-3016; U1111-1252-6589 (Other: WHO Universal Trial Number)
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2023-10

CONDITIONS: Pouchitis; Irritable Pouch Syndrome
MeSH Terms: conditions — Pouchitis | interventions — Liraglutide; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, 2-period, placebo-controlled, crossover proof of concept study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liraglutide then Placebo (Experimental): Participants will be randomly assigned to 6-week Liraglutide treatment. Then after a 5-day washout, treatment will continue with 6 weeks of placebo.
  Interventions: Drug: Liraglutide Pen Injector; Drug: Placebo Pen Injector
- Placebo then Liraglutide (Experimental): Participants will be randomly assigned to 6-week placebo treatment. Then after a 5-day washout, treatment will continue with 6 weeks of Liraglutide.
  Interventions: Drug: Liraglutide Pen Injector; Drug: Placebo Pen Injector

INTERVENTIONS:
Drug: Liraglutide Pen Injector — Treatment will be initiated at 0.6 mg per day for one week. The patient will be instructed to increase the dose to 1.2/day and 1.8 mg /day in week 2 and in week 3, respectively. From week 3 after the start of the drug until week 6 the patient will apply 1.8 mg/day liraglutide. In case of intolerance (e.g. occurrence of refractory nausea) at a higher dose (e.g. 1.8 mg daily, the highest dose in this trial) liraglutide can be reduced to the previous level.
  Other Names: Victoza
Drug: Placebo Pen Injector — Matching placebo pens used to administer normal saline in the same fashion as for liraglutide
  Other Names: Saline

SUMMARY:
Patients with an ileal pouch-anal anastomosis(IPAA; pouch) due to refractory inflammatory bowel disease and increased bowel frequency in the absence of significant pouch inflammation will be randomized to liraglutide or placebo in a prospective cross over study.

DETAILED DESCRIPTION:
Randomized, double-blind, 2-period, placebo- controlled, crossover proof of concept study.

Ten patients with increased bowel frequency defined as bowel frequency > 8 bowel movements in 24 hours on at least 4 of 7 days/week and presence of high bowel frequency > 4 weeks despite adequate therapy for acute pouchitis or Crohn's like disease of the pouch will be randomized to either liraglutide or placebo treatment for 6 weeks (Period 1). Subjects will be randomized 1:1 to 1 of 2 treatment sequences, liraglutide-placebo or placebo-liraglutide, and receive either liraglutide or volume-matched placebo. After a wash-out period of at least 5 days (the half-life of liraglutide is 11-12 hours, thus the minimal washout period of 5 days is equal to 10 half-life's) patients will be crossed over to the other treatment arm (Period 2). Since high bowel frequency can result in significant malaise and dehydration, patients not responding to the respective therapies in period 1 may be crossed over after 4 weeks of therapy or in period 2 can be terminated early at week 4. The rationale behind the early termination is based on 2 open-label cohorts reporting the efficacy of liraglutide or exenatide in patients with high output ileostomies (the patient group the most comparable to the pouch patient population). Glucagon-like peptide- 1 (GLP-1) receptor agonist therapy even at the lowest dose showed an almost immediate effect reducing the ostomy output after 1-3 days in most patients.Thus, patients not responding to a 4-week therapy with a GLP-1receptor agonist are highly unlikely to respond if the therapy would be continued.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained before any trial-related procedures
* Age > 18 years
* Patients with IPAA and bowel frequency > 8 bowel movements in 24 hours on at least 4 of 7 days/week and presence of high bowel frequency > 4 weeks despite adequate therapy for acute pouchitis or Crohn's like disease of the pouch

Exclusion Criteria:

* Significant pouch inflammation defined as an endoscopic pouch disease activity index (PDAI ) ≥ 4
* Known stricture of the ileo-anal anastomosis or afferent limb stricture
* New onset of high bowel frequency in the setting of acute pouchitis
* IPAA since < 6 months
* Known Clostridium difficile pouchitis
* Known clinically significant chronic nausea and/or vomiting in the past
* Known type 1 or type 2 diabetes
* History of or active neoplasia
* Personal or family history of medullary thyroid carcinoma or Multiple Endocrine Neoplasia syndrome type 2
* Renal impairment defined as glomerular filtration rate (glomerular filtration rate < 30)
* Clinically significant decompensated liver disease defined as elevation of aspartate aminotransferase , alanine transaminase or bilirubin > 2-fold the upper limits of normal (Primary Sclerosing Cholangitis with liver function tests (LFT's) <1.5 upper limits of normal can be included)
* New York Heart Association class 3 or greater heart failure or recent (within 6 months) cardiovascular event
* Prior history of pancreatitis
* Prior treatment with a GLP-1receptor agonist
* Known hypersensitivity to liraglutide or any product components
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method.
* Participation in any clinical trial of an approved or non-approved investigational medicinal product within 30 days before screening.
* Any disorder, which in the investigator's opinion might jeopardize patient's safety or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Herfarth, MD, PhD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 3 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina [UNC].
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Result] Herfarth H, Long MD, Hansen JJ, Anderson C, English E, Buse JB, Barnes EL. Efficacy and Safety of Liraglutide in Patients With an Ileal Pouch-Anal Anastomosis and Chronic High Bowel Frequency: A Placebo-Controlled, Crossover, Proof-of-Concept Study. Am J Gastroenterol. 2024 Sep 1;119(9):1935-1938. doi: 10.14309/ajg.0000000000002801. Epub 2024 Apr 12. PMID 38668926

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to an interruption in drug supply, the study was terminated after 8 of 10 patients were included.
Groups:
- Liraglutide Then Placebo: Participants first received Liraglutide treatment for 6 weeks. After a 5-day washout, they then received Placebo treatment for 6 weeks.
  Liraglutide Pen Injector: Treatment will be initiated at 0.6 mg per day for one week. The patient will be instructed to increase the dose to 1.2/day and 1.8 mg /day in week 2 and in week 3, respectively. From week 3 after the start of the drug until week 6 the patient will apply 1.8 mg/day liraglutide. In case of intolerance (e.g. occurrence of refractory nausea) at a higher dose (e.g. 1.8 mg daily, the highest dose in this trial) liraglutide can be reduced to the previous level.
  Placebo Pen Injector: Matching placebo pens used to administer normal saline in the same fashion as for liraglutide
- Placebo Then Liraglutide: Participants first received Placebo treatment for 6 weeks. After a 5-day washout, they then received Liraglutide treatment for 6 weeks.
  Liraglutide Pen Injector: Treatment will be initiated at 0.6 mg per day for one week. The patient will be instructed to increase the dose to 1.2/day and 1.8 mg /day in week 2 and in week 3, respectively. From week 3 after the start of the drug until week 6 the patient will apply 1.8 mg/day liraglutide. In case of intolerance (e.g. occurrence of refractory nausea) at a higher dose (e.g. 1.8 mg daily, the highest dose in this trial) liraglutide can be reduced to the previous level.
  Placebo Pen Injector: Matching placebo pens used to administer normal saline in the same fashion as for liraglutide
Period: First Intervention
Arm/Group | Liraglutide Then Placebo | Placebo Then Liraglutide
Started | 3 | 5
Completed | 3 | 5
Not Completed | 0 | 0
Period: Washout
Arm/Group | Liraglutide Then Placebo | Placebo Then Liraglutide
Started | 3 | 5
Completed | 3 | 5
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Liraglutide Then Placebo | Placebo Then Liraglutide
Started | 3 | 5
Completed | 3 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide Then Placebo | Placebo Then Liraglutide | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 49 [42 to 55] | 52 [44 to 65] | 51 [42 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 5 | 8
Daily bowel frequency [Mean (Standard Deviation); unit: bowel movements/day] — Data collected using participant diaries.
  bowel movements/day | 10.9 (2.1) | 12.8 (2.0) | 12.1 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean % Reduction of Bowel Frequency in Percent of the Mean 7-day Bowel Frequency After 4 Weeks of Therapy on Liraglutide vs Placebo Compared to Baseline .
Description: Mean percentage reduction of 7-day bowel frequency after 4 weeks of therapy on Liraglutide vs placebo compared to baseline (baseline is defined as the mean 7-day bowel frequency in a 7-day period during the screening period before week 0).
  Due to the cross-over design, the outcome is reported depending on randomization in treatment period 1 at week 4 and treatment period 2 at week 10 vs baseline.
Time Frame: Baseline, Week 4 (treatment period 1) and week 10 (treatment period 2)
Population: Analyses were performed according to treatment with Liraglutide vs Placebo (not according to arm/sequence).
Measure: Mean (Standard Deviation); unit: percentage reduction of bowel frequency
Groups:
- Liraglutide: 6-week Liraglutide treatment. Liraglutide Pen Injector: Treatment will be initiated at 0.6 mg per day for one week. The patient will be instructed to increase the dose to 1.2/day and 1.8 mg /day in week 2 and in week 3, respectively. From week 3 after the start of the drug until week 6 the patient will apply 1.8 mg/day liraglutide. In case of intolerance (e.g. occurrence of refractory nausea) at a higher dose (e.g. 1.8 mg daily, the highest dose in this trial) liraglutide can be reduced to the previous level.
- Placebo: 6-week placebo treatment. Placebo Pen Injector: Matching placebo pens used to administer normal saline in the same fashion as for liraglutide
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 8 | 8
percentage reduction of bowel frequency | 36.3 (19.8) | 17.3 (15.7)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; The 2 treatment modalities, Liraglutide and Placebo, were compared. A repeated-measures mixed model was fitted to the data, with treatment (liraglutide or placebo), period, and treatment sequence as fixed effects and the repeated measures within the subject as a random effect; Test type: Superiority; p < 0.03, Mixed Models Analysis — A priori threshold for significance was < 0.05. Significance level liraglutide vs. placebo in percent reduction of bowel frequency at week 4 vs. baseline

2. Secondary Outcome: Change in the 7 Day Mean Number of Day and Night Bowel Frequency at Week 4 and 6 vs Baseline on Liraglutide vs Placebo
Description: Bowel frequency during the day and night was recorded on a daily basis. The 7-day mean number of bowel movements during the day (from getting up until bedtime) and during the night (during sleep) at baseline and at weeks 4 and 6 on liraglutide or placebo therapy is depicted.
  Baseline, week 4 and week 6 (treatment period 1) and week 10 and week 12 (treatment period 2)
Time Frame: Baseline, Week 4 and week 6 (treatment period 1) and week 10 and week 12 (treatment period 2)
Population: Analyses were performed according to treatment with Liraglutide vs Placebo (not according to arm/sequence).
Measure: Mean (Standard Deviation); unit: Bowel movements / day or night
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 8 | 8
Bowel movements / day or night
  Baseline Bowel Frequency Day | 8.8 (2.3) | 8.8 (2.3)
  Baseline Bowel Frequency Night | 3.3 (1.7) | 8.8 (2.3)
  Week 4 Day | 5.3 (2.2) | 6.9 (2.2)
  Week 4 Night | 2.3 (1.1) | 3.1 (1.6)
  Week 6 Day | 5.4 (1.9) | 7.0 (2.0)
  Week 6 Night Placebo week 6 | 2.1 (1.0) | 3.1 (1.8)

3. Secondary Outcome: Discontinuation of Therapy in Each Treatment Arm
Description: Number of patients discontinuing Liraglutide therapy in treatment or placebo arm due to intolerance in treatment period 1 before week 6 or treatment period 2 before week 12
Time Frame: treatment period 1 before week 6 or treatment period 2 before week 12
Population: Analyses were performed according to treatment with Liraglutide vs Placebo (not according to arm/sequence).
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

4. Secondary Outcome: Mean % Reduction of Bowel Frequency in Percent of the Mean 7-day Bowel Frequency After 6 Weeks of Therapy on Liraglutide vs Placebo Compared to Baseline.
Description: Mean percentage reduction of 7-day bowel frequency after 6 weeks of therapy on Liraglutide vs placebo compared to baseline (baseline is defined as the mean 7-day bowel frequency in a 7-day period during the screening period before week 0).
  Due to the cross-over design, the outcome is reported depending on randomization in treatment period 1 at week 6 or treatment period 2 at week 12 vs baseline.
Time Frame: Baseline, week 6 (treatment period 1) and week 12 (treatment period 2)
Population: Analyses were performed according to treatment with Liraglutide vs Placebo (not according to arm/sequence).
Measure: Mean (Standard Deviation); unit: Percent reduction of bowel frequency
Groups:
- Liraglutide: Mean reduction of bowel frequency in percent of the mean 7-day bowel frequency after 6 weeks of therapy on Liraglutide compared to baseline
- Placebo: Mean reduction of bowel frequency in percent of the mean 7-day bowel frequency after 6 weeks of therapy on Placebo compared to baseline
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 8 | 8
Percent reduction of bowel frequency | 36.8 (18.7) | 15.7 (5.3)
Statistical Analysis 1: Comparison: Liraglutide vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.01, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: The adverse events were collected from each study participant from the screening visit until the last study visit at week 14
Arm/Group | Liraglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=8) | Placebo (N=8)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Diarrhea (intermittent) (Gastrointestinal disorders) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Fatigue (General disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Acid reflux (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hypoglycemic episode (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Hair loss (General disorders) | 1 (1) | 0 (0)
Chest tightness (General disorders) | 1 (1) | 0 (0)
Index finger n numbness (Nervous system disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hiccup (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small cross-over proof of concept study. The findings need to be verified in a more extensive prospective randomized study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT04763564/Prot_SAP_000.pdf